CLINICAL TRIAL: NCT00713284
Title: A Pilot Study to Evaluate the Safety and Efficacy of Mycophenolate Sodium (Myfortic®) in Combination With Sirolimus (Rapamune®) in Stable Renal Allograft Recipients
Brief Title: Study Evaluating Conversion From Tacrolimus to Sirolimus in Stable Kidney Transplant Recipients Receiving Myfortic
Acronym: MYFIIRP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: California Pacific Medical Center Research Institute (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, V. Ram Peddi, Medical Doctor, California Pacific Medical Center Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KTXP_US28_MYFIIRP07
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-08

CONDITIONS: Renal Transplantation
Keywords: Kidney transplantation; Sirolimus; Immunosuppression; Tacrolimus
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study (Other): All subjects who enroll in this study will be converted from their calcineurin inhibitor to sirolimus. There is no comparotor arm
  Interventions: Drug: sirolimus

INTERVENTIONS:
Drug: sirolimus — Oral tablet(s) taken daily for 6 months; dose will be based on serum trough levels.
  Other Names: Rapamune; rapamycin

SUMMARY:
The purpose of this study is to determine whether the combination of Myfortic and sirolimus is effective at preventing rejection while preserving kidney function in stable kidney transplant recipients.

DETAILED DESCRIPTION:
One-year graft survival after renal transplantation dramatically improved with the addition of calcineurin inhibitors (tacrolimus or cyclosporine) to maintenance immunosuppression regimens. Much of this improvement in early graft survival has been attributed to the efficacy of the calcineurin inhibitors in preventing early acute rejection episodes. However, long-term graft survival has not improved to as great of a magnitude as the improvements in short-term survival. In addition, research shows progressive decline in kidney function throughout the years post-transplantation. Clinical research now focuses on improving long term graft survival while maintaining long-term kidney function.

The leading cause of graft loss has been attributed to chronic allograft nephropathy (CAN). Risk factors for CAN include: prolonged ischemia time, delayed graft function, acute rejection episodes and calcineurin inhibitor nephrotoxicity (CIN). CIN has been identified as the most common identifiable contributor to CAN and the chief cause of late histologic injury and ongoing decline in renal function. At 10 years post-transplant, CIN has been found to be universally prevalent.

Calcineurin inhibitor minimization and elimination studies have sought to improve long-term allograft function by minimizing exposure to these nephrotoxic agents. Studies have demonstrated that early withdrawal of cyclosporine from a cyclosporine, sirolimus and steroid immunosuppression regimen at 3 months post-transplant improved renal function and graft survival at 48 months post-transplant. Other studies have demonstrated diminished prevalence of CAN at 2 years post-transplant in those patients maintained on sirolimus as compared with cyclosporine. Kidney function was also significantly improved with lower serum creatinine and higher GFR in the sirolimus maintenance group.

Sirolimus is a macrolide antibiotic immunosuppressive agent that exerts its mechanism of action by inhibiting the mTOR signaling cascade. In clinical trials, sirolimus was found to lack nephrotoxic effects when compared to cyclosporine. In kidney transplantation, multiple studies have demonstrated safety and efficacy of sirolimus in calcineurin inhibitor avoidance and withdrawal protocols.

Myfortic® (mycophenolate acid) is an enteric coated formulation of mycophenolic acid (MPA) approved for the prevention of rejection in kidney transplant recipients in combination with cyclosporine and corticosteroids. Myfortic® has no documented nephrotoxic effects. Mycophenolate mofetil (MMF), a prodrug of MPA also does not demonstrate nephrotoxic effects. Early studies have demonstrated therapeutic equivalence between Myfortic® and MMF both in de novo renal transplants and in conversion studies where MMF is converted to Myfortic at least 6 months after renal transplantation. Thus, studies demonstrating safety and efficacy of MMF with sirolimus in calcineurin inhibitor withdrawal protocols should also hold true using Myfortic® in such regimen.

This study will assess the safety and efficacy of Myfortic® when used in a simultaneous sirolimus conversion and calcineurin inhibitor withdrawal regimen in stable renal transplant recipients. Study subjects will receive immunosuppression consisting of Myfortic®, tacrolimus and corticosteroids (prednisone) starting the day of transplant. Conversion from tacrolimus (Prograf) to sirolimus (Rapamune) will occur between 90 and 180 days post cadaver-donor or living-donor renal transplant. All participants will be converted from tacrolimus to sirolimus and remain on Myfortic® and their current corticosteroid taper.

ELIGIBILITY:
Inclusion Criteria I (-1 to 7 days post renal allograft transplant):

* Male or female patient 18 years of age or older.
* Patient has been fully informed of study procedures and requirements, has signed an IRB approved consent form and is willing and able to follow study procedures.

Exclusion Criteria I (-1 to 7 days post renal allograft transplant):

* Patient has previously received an organ transplant.
* Patient has an identified donor specific antibody prior to transplant
* Patient is known to be seropositive for the human immunodeficiency virus (HIV).
* Patient has active Hepatitis C or B infection documented by a positive DNA PCR. Patients who are seropositive for Hepatitis C virus (HCV) or B virus (HBV) but have negative HCV-RNA or HBV-DNA by PCR may be included.
* Patient has a current malignancy or a history of malignancy within the past 5 years, except non-metastatic basal or squamous cell carcinoma of the skin that has been treated successfully.
* Patient has an uncontrolled infection or unstable medical condition that could interfere with the study objectives.
* Patient is currently taking or has been taking an investigational drug in the past 30 days.
* Patient has a known hypersensitivity to sirolimus or Myfortic®.
* Patient is pregnant or lactating.
* Patient is unlikely to comply with the visits scheduled in the protocol.
* Patient has any form of substance abuse, psychiatric disorder or a condition that, in the opinion of the investigator, may invalidate communication with the investigator.

Inclusion Criteria II (90 - 180 days post renal allograft transplant):

* Patient is 90 to 180 days after having received a primary living- or cadaver-donor renal allograft
* Patient has been maintained on a regimen of tacrolimus, Myfortic® and corticosteroids prior to study enrollment.
* Patient has a stable allograft defined as calculated GFR > 30 mL/min using Nankivell equation.
* Patient has been fully informed of study procedures and requirements, has signed an IRB approved consent form and is willing and able to follow study requirements.
* Female patients of child bearing potential must use at least one reliable form of contraception unless they are status post bilateral tubal ligation, bilateral oophorectomy or hysterectomy. Effective contraception must be used for the duration of the study.

Exclusion Criteria II (90 - 180 days post renal allograft transplant):

* Patient has experienced an acute graft rejection of ≥ Banff '97 1b or humoral rejection as determined by biopsy within the first 90 days post-transplant
* Patient has experienced an acute graft rejection of ≤ Banff 97 1a as determined by biopsy within 30 days prior to Baseline visit.
* Patient has untreated hypercholesterolemia defined as triglycerides > 300 or total cholesterol >200 within the previous 30 days.
* Patient is currently (< 7 days) leukopenic defined as WBC < 3,000 cells/mL or thrombocytopenic defined as platelets < 100,000 cells/mL.
* Patient has significant liver disease, defined as having during the past 30 days continuously elevated AST (SGOT) and/or ALT (SGPT) levels greater than 3 times the upper value of normal range.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: V. Ram Peddi, MD, Principal Investigator — California Pacific Medical Center
Locations (1):
- California Pacific Medical Center; Barry S. Levin, MD Department of Transplantation, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
No data will be shared with other researchers

REFERENCES:
- [Background] Merion RM, White DJ, Thiru S, Evans DB, Calne RY. Cyclosporine: five years' experience in cadaveric renal transplantation. N Engl J Med. 1984 Jan 19;310(3):148-54. doi: 10.1056/NEJM198401193100303. PMID 6361559
- [Background] Pirsch JD, Miller J, Deierhoi MH, Vincenti F, Filo RS. A comparison of tacrolimus (FK506) and cyclosporine for immunosuppression after cadaveric renal transplantation. FK506 Kidney Transplant Study Group. Transplantation. 1997 Apr 15;63(7):977-83. doi: 10.1097/00007890-199704150-00013. PMID 9112351
- [Background] Nankivell BJ, Borrows RJ, Fung CL, O'Connell PJ, Allen RD, Chapman JR. The natural history of chronic allograft nephropathy. N Engl J Med. 2003 Dec 11;349(24):2326-33. doi: 10.1056/NEJMoa020009. PMID 14668458
- [Background] Hariharan S, McBride MA, Cherikh WS, Tolleris CB, Bresnahan BA, Johnson CP. Post-transplant renal function in the first year predicts long-term kidney transplant survival. Kidney Int. 2002 Jul;62(1):311-8. doi: 10.1046/j.1523-1755.2002.00424.x. PMID 12081593
- [Background] Oberbauer R, Segoloni G, Campistol JM, Kreis H, Mota A, Lawen J, Russ G, Grinyo JM, Stallone G, Hartmann A, Pinto JR, Chapman J, Burke JT, Brault Y, Neylan JF; Rapamune Maintenance Regimen Study Group. Early cyclosporine withdrawal from a sirolimus-based regimen results in better renal allograft survival and renal function at 48 months after transplantation. Transpl Int. 2005 Jan;18(1):22-8. doi: 10.1111/j.1432-2277.2004.00052.x. PMID 15612979
- [Background] Flechner SM, Kurian SM, Solez K, Cook DJ, Burke JT, Rollin H, Hammond JA, Whisenant T, Lanigan CM, Head SR, Salomon DR. De novo kidney transplantation without use of calcineurin inhibitors preserves renal structure and function at two years. Am J Transplant. 2004 Nov;4(11):1776-85. doi: 10.1111/j.1600-6143.2004.00627.x. PMID 15476476
- [Background] Stallone G, Di Paolo S, Schena A, Infante B, Grandaliano G, Battaglia M, Gesualdo L, Schena FP. Early withdrawal of cyclosporine A improves 1-year kidney graft structure and function in sirolimus-treated patients. Transplantation. 2003 Apr 15;75(7):998-1003. doi: 10.1097/01.TP.0000057240.95073.35. PMID 12698087
- [Background] Mota A, Arias M, Taskinen EI, Paavonen T, Brault Y, Legendre C, Claesson K, Castagneto M, Campistol JM, Hutchison B, Burke JT, Yilmaz S, Hayry P, Neylan JF; Rapamune Maintenance Regimen Trial. Sirolimus-based therapy following early cyclosporine withdrawal provides significantly improved renal histology and function at 3 years. Am J Transplant. 2004 Jun;4(6):953-61. doi: 10.1111/j.1600-6143.2004.00446.x. PMID 15147430
- [Background] Morales JM, Wramner L, Kreis H, Durand D, Campistol JM, Andres A, Arenas J, Negre E, Burke JT, Groth CG; Sirolimus European Renal Transplant Study Group. Sirolimus does not exhibit nephrotoxicity compared to cyclosporine in renal transplant recipients. Am J Transplant. 2002 May;2(5):436-42. doi: 10.1034/j.1600-6143.2002.20507.x. PMID 12123209
- [Background] Reitamo S, Spuls P, Sassolas B, Lahfa M, Claudy A, Griffiths CE; Sirolimus European Psoriasis Study Group. Efficacy of sirolimus (rapamycin) administered concomitantly with a subtherapeutic dose of cyclosporin in the treatment of severe psoriasis: a randomized controlled trial. Br J Dermatol. 2001 Sep;145(3):438-45. doi: 10.1046/j.1365-2133.2001.04376.x. PMID 11531834
- [Background] Flechner SM, Goldfarb D, Modlin C, Feng J, Krishnamurthi V, Mastroianni B, Savas K, Cook DJ, Novick AC. Kidney transplantation without calcineurin inhibitor drugs: a prospective, randomized trial of sirolimus versus cyclosporine. Transplantation. 2002 Oct 27;74(8):1070-6. doi: 10.1097/00007890-200210270-00002. PMID 12438948
- [Background] Simmons WD, Rayhill SC, Sollinger HW. Preliminary risk-benefit assessment of mycophenolate mofetil in transplant rejection. Drug Saf. 1997 Aug;17(2):75-92. doi: 10.2165/00002018-199717020-00001. PMID 9285199
- [Background] Budde K, Curtis J, Knoll G, Chan L, Neumayer HH, Seifu Y, Hall M; ERL B302 Study Group. Enteric-coated mycophenolate sodium can be safely administered in maintenance renal transplant patients: results of a 1-year study. Am J Transplant. 2004 Feb;4(2):237-43. doi: 10.1046/j.1600-6143.2003.00321.x. PMID 14974945
- [Background] Salvadori M, Holzer H, de Mattos A, Sollinger H, Arns W, Oppenheimer F, Maca J, Hall M; ERL B301 Study Groups. Enteric-coated mycophenolate sodium is therapeutically equivalent to mycophenolate mofetil in de novo renal transplant patients. Am J Transplant. 2004 Feb;4(2):231-6. doi: 10.1046/j.1600-6143.2003.00337.x. PMID 14974944

RESULTS

PARTICIPANT FLOW:
Groups:
- Sirolimus Conversion: All subjects who enroll in this study will be converted from their calcineurin inhibitor to sirolimus.
Period: Overall Study
Arm/Group | Sirolimus Conversion
Started | 29 (29 participants were screened but only 13 eligible for conversion and continue in the study.)
Completed | 13
Not Completed | 16

BASELINE CHARACTERISTICS:
Arm/Group | Sirolimus Conversion
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.15 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 13
Transplant Type [Count of Participants; unit: Participants]
  Deceased donor | 6
  Living Unrelated donor | 4
  Living Related donor | 3
Expanded Criteria Donor [Count of Participants; unit: Participants]
  Expanded Criteria Donor | 2
  Not Expanded Criteria Donor | 11
Time to Conversion [Mean (Standard Deviation); unit: days] | 147.85 (36)

OUTCOME MEASURES:

1. Primary Outcome: Renal Allograft Function
Description: Renal allograft function will be assessed based on serum creatinine
Time Frame: six months
Population: One patient experienced an adverse drug reaction and was withdrawn from study treatment one month after conversion
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sirolimus Conversion
Number analyzed (Participants) | 13
mg/dL
  Creatinine (Baseline) | 1.34 (0.24)
  Creatinine (6 months): number analyzed (Participants) | 12
  Creatinine (6 months) | 1.38 (0.31)
Statistical Analysis 1: Comparison: Sirolimus Conversion; Test type: Other; p < 0.05, t-test, 1 sided

ADVERSE EVENTS:
Arm/Group | Sirolimus Conversion
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 1/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus Conversion (N=13)
Rise in creatinine (Renal and urinary disorders) | 1 (1)
Edema (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitation is small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No